CLINICAL TRIAL: NCT05708729
Title: Neuromodulation for Central Post-stroke Pain: Mechanism, Safety and Outcome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S66772; CIV-22-09-040829 (Other: FAMHP)
Record Dates: First submitted 2023-01-09; First posted 2023-02-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Central Post-stroke Pain; CPSP
Keywords: neuromodulation; DBS; rTMS; MCS

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding for rTMS (active stimulation vs sham stimulation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patients with CPSP which is pharmacorefractory and have a good analgesic response to M1-rTMS (Experimental): Diagnosed with definite CPSP (Treede-Klit criteria), which is pharmacorefractory (i.e. amitriptyline 75mg/d 4w, lamotrigine 200mg/d 8w and pregabalin 600mg/d resulting in <50% VAS reduction and/or intolerable side-effects).
  A good analgesic response to M1-rTMS is defined as: ≥50% mean 10-d VAS reduction immediately following vs. before active M1-rTMS minus mean 10-d VAS reduction immediately following vs. pre sham M1-rTMS. A good analgesic response gives a high positive predictive value for pain reduction by MCS.
  Interventions: Device: MCS surgery for CPSP
- Patients with CPSP which is pharmacorefractory with less analgesic M1-rTMS response (Experimental): Diagnosed with definite CPSP (Treede-Klit criteria), which is pharmacorefractory (i.e. amitriptyline 75mg/d 4w, lamotrigine 200mg/d 8w and pregabalin 600mg/d resulting in <50% VAS reduction and/or intolerable side-effects).
  Patients with less analgesic M1-rTMS response (n≈20) will be 1:1 randomized to either MCS (≈10) or Vc-DBS (n≈10).
  Interventions: Device: MCS surgery for CPSP; Device: Vc-DBS surgery for CPSP

INTERVENTIONS:
Device: MCS surgery for CPSP — The investigational devices that will be used for the MCS surgeries are the following: the Vanta with AdaptiveStim Technology Primary cell neurostimulator or the Intellis Implantable Neurostimulator with AdaptiveStim Technology from Medtronic, Inc. (MN, USA). These implantable neurostimulators are intended to generate electrical pulses and to deliver stimulation trough one or more leads as part of a neurostimulation system for pain therapy in adults.
Device: Vc-DBS surgery for CPSP — For the deep brain stimulation procedure, we will use Vercise stimulators from Boston Scientific together with the Cartesia Directional Leads or the Percept PC stimulator from Medtronic.
  Arms: Patients with CPSP which is pharmacorefractory with less analgesic M1-rTMS response

SUMMARY:
Central post-stroke pain (CPSP) is an often pharmacorefractory type of neuropathic pain that develops in 8% of stroke patients. CPSP has been treated with three distinct types of neuromodulation (deep brain stimulation of the sensory thalamus (Vc-DBS), motor cortex repetitive transcranial magnetic stimulation (M1-rTMS), and motor cortex stimulation (MCS)), but the level of evidence for these procedures is very low. Moreover, data on the changes in pain brain circuitry in CPSP, and the effect of neuromodulation on this circuitry is very limited.

DETAILED DESCRIPTION:
In this project, we propose a prospective double-blind randomized crossover on/off study in 32 CPSP patients. These patients will undergo M1-rTMS and either MCS or Vc-DBS. Before and after active and inactive stimulation they will be assessed with clinical scales for pain, function, quality of life and depression. Adverse events will be monitored. This allows to measure the outcome and safety of neuromodulation in CPSP.

In addition, we will have functional magnetic resonance imaging (fMRI) and positron emission tomography (PET) use. This will provide insight into the pathological changes in the pain circuitry, and the influence of neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide voluntary written informed consent of the participant prior to any screening procedures
2. Male or female patients
3. Aged 18-70 years
4. Diagnosed with definite CPSP (Treede-Klit criteria) (1, 9), which is pharmacorefractory (i.e. amitriptyline 75mg/d 4w, lamotrigine 200mg/d 8w and pregabalin 600mg/d resulting in <50% VAS reduction and/or intolerable side-effects)

Exclusion Criteria:

1. Aphasia
2. Pregnancy or intention to become pregnant in the following year
3. Medical inoperability
4. Impossibility to temporarily withhold anticoagulation or anti-platelet medication
5. Impossibility to undergo MRI, fMRI and/or PET imaging
6. Complete destruction of the stimulation target region (M1 or Vc)
7. Uncontrolled seizures
8. Expected relocation in the following year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The relative difference in pain intensity (Visual Analogue Scale; VAS) immediately following 10 sessions of active vs. inactive rTMS; | After completion of all rTMS sessions (approximately one month before surgery)
  The patients will receive 10 sessions (1/d) of active and 10 sessions (1/d) of sham M1-rTMS with a 8-week wash-out period in between.
The relative difference in pain intensity (Visual Analogue Scale; VAS) immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS. | After completion of the 4 weeks of active vs. inactive MCS or Vc-DBS (approximately at 9 months after surgery)
  Stimulation will be optimised for all patients up to 5 months post-surgery (Vc-DBS or MCS). After 2 weeks of wash-out, active and inactive stimulation will be offered in a double-blinded fashion for 4 weeks, with 2 weeks of wash-out in between.

SECONDARY OUTCOMES:
The relative difference in pain symptoms* immediately following 10 sessions of active vs. inactive rTMS; | Immediately after completion of the 10 sessions of active (1 per day, on 10 consecutive days) and 10 sessions of sham (1 per day, on 10 consecutive days) M1-rTMS with a 8 weeks washout period inbetween
  * as measured through the Neuropathic Pain Symptom Inventory (NPSI) and Patient Global Impression of Change (PGIC)
The relative difference in use of analgesics* immediately following 10 sessions of active vs. inactive rTMS; | Immediately after completion of the 10 sessions of active (1 per day, on 10 consecutive days) and 10 sessions of sham (1 per day, on 10 consecutive days) M1-rTMS with a 8 weeks washout period inbetween
  * as measured through the Medication Quantification Scale
The relative difference in functionality* immediately following 10 sessions of active vs. inactive rTMS; | Immediately after completion of the 10 sessions of active (1 per day, on 10 consecutive days) and 10 sessions of sham (1 per day, on 10 consecutive days) M1-rTMS with a 8 weeks washout period inbetween
  * as measured through the Functional Independence Measure (FIM)
The relative difference in quality of life* immediately following 10 sessions of active vs. inactive rTMS; | Immediately after completion of the 10 sessions of active (1 per day, on 10 consecutive days) and 10 sessions of sham (1 per day, on 10 consecutive days) M1-rTMS with a 8 weeks washout period inbetween
  * as measured through the 36-Item Short-Form Health Survey (SF-36 QoLS)
The relative difference in mood* immediately following 10 sessions of active vs. inactive rTMS; | Immediately after completion of the 10 sessions of active (1 per day, on 10 consecutive days) and 10 sessions of sham (1 per day, on 10 consecutive days) M1-rTMS with a 8 weeks washout period inbetween
  * as measured through the Beck Depression Inventory (BDI)
The relative difference in pain symptoms* immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS; | immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  * as measured through the Neuropathic Pain Symptom Inventory (NPSI) and Patient Global Impression of Change (PGIC)
The relative difference in use of analgesics* immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS; | immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  * as measured through the Medication Quantification Scale
The relative difference in functionality* immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS; | immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  * as measured through the Functional Independence Measure (FIM)
The relative difference in quality of life* immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS; | immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  * as measured through the 36-Item Short-Form Health Survey (SF-36 QoLS)
The relative difference in mood* immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS; | immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  * as measured through the Beck Depression Inventory (BDI)
The relative difference in metabolic activity (as measured through FDG-PET) in pain matrix areas immediately following 10 sessions of active vs. inactive rTMS; | Immediately after completion of the 10 sessions of active (1 per day, on 10 consecutive days) and 10 sessions of sham (1 per day, on 10 consecutive days) M1-rTMS with a 8 weeks washout period inbetween
The relative difference in metabolic activity (as measured through rsMRI) in pain matrix areas immediately following 10 sessions of active vs. inactive rTMS; | Immediately after completion of the 10 sessions of active (1 per day, on 10 consecutive days) and 10 sessions of sham (1 per day, on 10 consecutive days) M1-rTMS with a 8 weeks washout period inbetween
The relative difference in metabolic activity (as measured through FDG-PET) in pain matrix areas immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS; | immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
The relative difference in metabolic activity (as measured through rsMRI) in pain matrix areas immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS; | immediately following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
The spike rate in the presence or absence of noxious/innocuous sensory stimuli (selected through baseline QSM); | Intraoperative
  *as measured through the microelectrodes (Vc-DBS) and paddle electrodes (MCS)
The spectral power* in the presence or absence of noxious/innocuous sensory stimuli (selected through baseline QSM); | Intraoperative
  *as measured through the microelectrodes (Vc-DBS) and paddle electrodes (MCS)
Other neurophysiological parameters* in the presence or absence of noxious/innocuous sensory stimuli (selected through baseline QSM); | Intraoperative
  *as measured through the microelectrodes (Vc-DBS) and paddle electrodes (MCS)
The spike rate* in the presence and absence of noxious and innocuous sensory stimuli (selected through baseline QSM) | following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  *as measured postoperatively through the implanted electrodes
The spectral power* in the presence and absence of noxious and innocuous sensory stimuli (selected through baseline QSM) | following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  *as measured postoperatively through the implanted electrodes
Other neurophysiological parameters* in the presence and absence of noxious and innocuous sensory stimuli (selected through baseline QSM) | following 4 weeks of active (with optimized stimulation parameters) vs. inactive MCS or Vc-DBS;
  *as measured postoperatively through the implanted electrodes
The safety for every procedure and during active and inactive rTMS, MCS and/or Vc-DBS. | during procedure and during active and inactive rTMS, MCS and/or Vc-DBS.
  *as measured by the AEs and SAEs
The safety for every procedure | during procedure
  *as measured by the AEs and SAEs
The safety during active and inactive rTMS | during active and inactive rTMS
  *as measured by the AEs and SAEs
The safety during active and inactive MCS or Vc-DBS. | during active and inactive MCS or Vc-DBS.
  *as measured by the AEs and SAEs

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No